CLINICAL TRIAL: NCT00342758
Title: Early Life Factors and Respiratory Health in Mexico City Children
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902005; 02-E-N005
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-10-15

CONDITIONS: Respiratory Ilness
Keywords: Asthma; Wheeze; Environment; Diet; Infection
MeSH Terms: conditions — Asthma; Respiratory Sounds; Infections

SUMMARY:
Early life exposures now appear to be important in modulation of the immune response and tendency to develop asthma. We plan to enroll a cohort of children at birth to study early life factors in the development of wheezing and respiratory illness during the first six years of life in Mexico City. In particular, we will consider the role of early diet (particularly antioxidant intake, lactation and obesity), infections, dust mite and cockroach antigens, traffic related air pollution, and environmental tobacco smoke. We will also consider the potential modifying effect of genetic predisposition with respect to the exposures of interest.

Approximately 6,800 children will be enrolled at birth. The goal is to follow the cohort though age 6. To increase the number of expected cases of asthma, we will partially enrich the cohort for increased risk of asthma by virtue of having a parent with doctor diagnosis of asthma or allergies; the remaining cohort will not be enriched to preserve generalizability.

Pregnant women enrolled in a prepaid health plan in Mexico City (the Insituto Mexicano de Seguridad Social, henceforth referred to as IMSS) will be screened for the study and invited to enrolled their newborns when they come for delivery at one of two IMSS hospitals. An initial home visit during the first three months of life will include assessment of environmental exposures and infant diet. Children will be followed through age six with yearly home visits, monitoring of acute lower respiratory illness during the first year of life and periodic review of the IMSS medical records.

We have chosen Mexico City because of the relatively low rates of asthma in the face of prevalent exposures to factors that are thought to increase asthma risk in urban areas in the United States. These include dust mites, cockroach, airborne pollutants and social factors such as low income and young maternal age. This pattern suggests that protective factors may be operating in Mexico City that could shed light on the etiology of worldwide childhood asthma epidemic. Potential candidates include exposure to certain early infections that shift the developing immune system away from the pattern of allergic asthmatic response. We are also especially interested in potential protective effects of early nutrition. Exposure to ozone in this population is the highest in North American and thus antioxidant intake may be especially important. In order to evaluate these protective hypotheses, we will also collect information on risk factors believed to be related to increased risk of asthma in US cities such as allergens, traffic related air pollutants, and lower respiratory infection with respiratory syncytial virus.

DETAILED DESCRIPTION:
Early life exposures now appear to be important in modulation of the immune response and tendency to develop asthma. We plan to enroll a cohort of children at birth to study early life factors in the development of wheezing and respiratory illness during the first six years of life in Mexico City. In particular, we will consider the role of early diet (particularly antioxidant intake, lactation and obesity), infections, dust mite and cockroach antigens, traffic related air pollution, and environmental tobacco smoke. We will also consider the potential modifying effect of genetic predisposition with respect to the exposures of interest.

Approximately 6,800 children will be enrolled at birth. The goal is to follow the cohort though age 6. To increase the number of expected cases of asthma, we will partially enrich the cohort for increased risk of asthma by virtue of having a parent with doctor diagnosis of asthma or allergies; the remaining cohort will not be enriched to preserve generalizability.

Pregnant women enrolled in a prepaid health plan in Mexico City (the Insituto Mexicano de Seguridad Social, henceforth referred to as IMSS) will be screened for the study and invited to enrolled their newborns when they come for delivery at one of two IMSS hospitals. An initial home visit during the first three months of life will include assessment of environmental exposures and infant diet. Children will be followed through age six with yearly home visits, monitoring of acute lower respiratory illness during the first year of life and periodic review of the IMSS medical records.

We have chosen Mexico City because of the relatively low rates of asthma in the face of prevalent exposures to factors that are thought to increase asthma risk in urban areas in the United States. These include dust mites, cockroach, airborne pollutants and social factors such as low income and young maternal age. This pattern suggests that protective factors may be operating in Mexico City that could shed light on the etiology of worldwide childhood asthma epidemic. Potential candidates include exposure to certain early infections that shift the developing immune system away from the pattern of allergic asthmatic response. We are also especially interested in potential protective effects of early nutrition. Exposure to ozone in this population is the highest in North American and thus antioxidant intake may be especially important. In order to evaluate these protective hypotheses, we will also collect information on risk factors believed to be related to increased risk of asthma in US cities such as allergens, traffic related air pollutants, and lower respiratory infection with respiratory syncytial virus.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must be pregnant coming to deliver.

Patients must have convenient access to a phone.

Patients must be residents of Mexico City, Mexico.

Women patients must not be planning to move from their current residence in the next two years or to drop their IMSS coverage .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6800
Dates: Start 2001-10-01; Study Completion 2007-10-15

CONTACTS AND LOCATIONS:
Locations (4):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States
- Mexico (3):
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Instituto Mexicano del Seguro Social, Mexico City
  - National Institute of Public Health, Mexico City